CLINICAL TRIAL: NCT05329207
Title: Effects of Web-Based Adolescent Health Promotion Program on Physical Activity, Nutrition and Mental Health in Hearing Impaired Adolescents
Brief Title: Effects of Web-Based Adolescent Health Promotion Program in Hearing Impaired Adolescents
Acronym: ASGE-FABES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hakan ORAKCI, PhD Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HAKAN ORAKCI PHD THESIS
Record Dates: First submitted 2022-01-19; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Health Promotion
Keywords: Hearing Impaired; Adolescent health; Health Promotion; Web-based; ASGE- FABES
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: The study was in the design type with pretest-posttest control group, repeated measures in randomized groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Intervention group) Hearing impaired adolescent experimental group (Experimental): Hearing Impaired Adolescent Group implemented Web-Based Adolescent Health Promotion Education Program
  Interventions: Behavioral: Experimental group
- (Control group) Hearing impaired adolescent control Group (No Intervention): Hearing Impaired Adolescent Group that did not apply Web-Based Adolescent Health Promotion Education Program

INTERVENTIONS:
Behavioral: Experimental group — Web Based Adolescent Health Promotion Education Program
  Other Names: ASGE-FABES
  Arms: (Intervention group) Hearing impaired adolescent experimental group

SUMMARY:
Our research is to evaluate the effect and applicability of the adolescent health promotion program, which includes multiple behavioral interventions, on physical activity, nutrition and mental health of hearing impaired adolescents living in the community.

DETAILED DESCRIPTION:
Purpose of the research; To evaluate the effect and applicability of the Web-Based Adolescent Health Promotion program, which includes multiple health behavior initiatives, on physical activity, nutrition, and stress management of hearing impaired adolescents in making healthy choices, assuming their own health responsibilities and acquiring healthy lifestyle behaviors.

Materials and methods; The research is a full experimental study with pretest-posttest control group, repeated measurement design, random groups.

Research sample; A total of 70 hearing-impaired adolescents aged 12-18, studying at Abdurrahman Gazi Sağlar Primary School, Van Special Education Vocational High School and Duyus Special Education and Rehabilitation Center affiliated to the Ministry of National Education in the city center of Van.

The data of the research; "Sociodemographic Characteristics Information Form", "Body Mass Index (BMI)", "Adolescent Nutrition Information Scale", "Adolescent Physical Activity Information Scale", "Adolescent Lifestyle Scale", "Adolescent Healthy Lifestyle Choices Scale", "Renewed Child" Anxiety and Depression Scale", "Daily Food Consumption Form", "Beverage Consumption Form", "Pedometer" were collected.

In the study; descriptive statistics will be evaluated with mean, standard deviation, percentage and frequency analysis. Comparisons between groups will be analyzed using Pearson's chi-square, Student's t-test, Mann Whitney-U test, Kruskal Wallis test, analysis of variance and Cohen's d effect size.

The results of this study;

* Physical Variables: Body Mass Index (BMI) and Weight
* Behavioral Variables: Weekly average number of steps and change, fruit and vegetable consumption amount, amount of water consumed, amount of sugary and acidic beverages consumed, "Adolescent Lifestyle" scale score average, "Adolescent" Lifestyle Choices scale score average,
* Cognitive Variables: "Adolescent Nutrition Knowledge" scale mean score, "Adolescent Physical Activity Knowledge" scale mean score, "Regenerated Child Anxiety and Depression" scale mean score will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impairment,
* In the 12-18 age group,
* Ability to access communication tools such as computers, tablets and smartphones and use the internet with these tools,
* Able to communicate in visual, sign language and written,
* Does not have a physical condition or disease that may prevent exercise,
* Volunteer to participate in the research,
* Permitted to participate in the research by their parents.

Exclusion Criteria:

* who want to withdraw from the research

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-10-18 (Estimated); Study Completion 2022-11-18 (Estimated)

PRIMARY OUTCOMES:
Physical Variables: | 9 months
  Body Mass Index (BMI- kg/m^2) and Weight (kg)

SECONDARY OUTCOMES:
Behavioral Variables: | 9 months
  The mean score of "Adolescent Lifestyle Scale" is used for behavioral change;
  * The scale requires a 4-point Likert-type response for each item. 1 for "Never", 2 for "Sometimes", 3 for "Often" and 4 for "Always"
  * The maximum score obtained from the scale is 160 and the minimum score is 40.
  * The scale does not have a cut-off point, as the score increases, the level of positive health behavior increases
Cognitive Variables 1: | 9 months
  The mean score of "Adolescent Nutrition Knowledge Scale" will be evaluated.
  Scoring
  1. Highlighted answer is correct
  2. Recode items
     1. If answer don't know (2), recode as no (0)
     2. If answer is correct, recode as (1)
     3. If answer is incorrect, recode as (0)
  3. After recoding, sum items 1-12
  4. Summed total will reflect the number of items answered correctly.
Cognitive Variables 2: | 9 months
  The mean score of "Adolescent Physical Activity Knowledge Scale" will be evaluated.
  Scoring
  1. Highlighted answer is correct
  2. Recode items
     1. If answer don't know (2), recode as no (0)
     2. If answer is correct, recode as (1)
     3. If answer is incorrect, recode as (0)
  3. After recoding, sum items 1-12
  4. Summed total will reflect the number of items answered correctly.
Cognitive Variables 3: | 9 months
  The mean score of "Regenerated Child Anxiety and Depression Scale" will be evaluated.
  The RCADS consists of 47 items developed to measure DSM-IV based symptoms of anxiety disorders and depression in children and adolescents.
  The subscales correspond to SAD (7 items), SP (9 items), GAD (6 items), PD (9 items), OCD (6 items), and MDD (10 items).
  It is scored on a 4-point scale (0 =never, 1 = sometimes, 2 = often, and 3 = always).

CONTACTS AND LOCATIONS:
Overall Officials: AYSUN ARDIÇ, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orakci H, Ardic A. The effect of web-based cope healthy lifestyles TEEN program on hearing-impaired adolescents: A randomized controlled trial. J Pediatr Nurs. 2025 Dec 18;86:590-602. doi: 10.1016/j.pedn.2025.12.006. Online ahead of print. PMID 41418421